CLINICAL TRIAL: NCT03029676
Title: The Assessment of Postoperative Cognitive Dysfunction After Transurethral Resection of Bladder Tumor Under Spinal Anesthesia
Brief Title: The Assessment of POCD After TURBT Under Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Karolina Dobrońska, MD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/1/2017
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Bladder Tumor; Postoperative Cognitive Dysfunction
Keywords: spinal anesthesia, TURBT, POCD, premedication
MeSH Terms: conditions — Urinary Bladder Neoplasms; Postoperative Cognitive Complications | interventions — Benzodiazepines; Midazolam; Analgesics, Opioid; Fentanyl; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Masking Description: the participant is not performed about the type of premedication performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Experimental): spinal anesthesia premedication with benzodiazepine and opioid
  Interventions: Drug: benzodiazepines; Drug: opioid; Procedure: spinal anesthesia
- Group K (Active Comparator): spinal anesthesia premedication with opioid
  Interventions: Drug: opioid; Procedure: spinal anesthesia

INTERVENTIONS:
Drug: benzodiazepines — sedative
  Other Names: midazolam
  Arms: Group B
Drug: opioid — analgetic, sedative
  Other Names: fentanyl
Procedure: spinal anesthesia

SUMMARY:
This study evaluates the influence of premedication on cognitive functions in patients undergoing transurethral resection of bladder tumor under spinal anesthesia. The aims of premedication are anxiolysis, analgesia and the reduction of perioperative risk among the patients with comorbidities. The patients will be randomly allocated to receive premedication either with opioid solely or with benzodiazepine combined with opioid. The anesthetic technique is standardized.

DETAILED DESCRIPTION:
Trans-urethral resection of bladder tumor (TURBT) is the basic endoscopic procedure for management of bladder cancer and if there are no contraindications, it is performed under spinal anesthesia. The condition usually occurs among elderly patients, every 9 of 10 is older than 55 years. At this age the postoperative cognitive dysfunction (POCD) is a common complication as the risk increases with age. There are some studies indicating that using benzodiazepines during the perioperative period can also increase the number of registered POCD in patients undergoing anesthesia. Postoperative cognitive dysfunction (POCD) occurs after operations under regional and general anesthesia as well. The study was planed to evaluate the risk of POCD among urological patients and to asses whether combining benzodiazepines with opioids for premedication increases this risk.

The participants after giving the informed consent can participate in the study. The Beck Depression Inventory is performed to rule out the patients with depression. The cognitive functions are tested with Montreal Cognitive Assessment before the surgery and subsequently in the first 24 hours after surgery, three weeks later (while patients come back to receive histopathological examination), and finally six months after surgery (during control cystoscopy).

During anesthesia, the patients will be randomly allocated to receive premedication either with opioid solely or with benzodiazepine combined with opioid. The anesthetic technique is standardized. If the premedication is needed before the surgery the hydroxyzine will be administrated.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* transurethral resection of the bladder tumor
* spinal anesthesia

Exclusion Criteria:

Exclusion Criteria:

* patients' refusal
* contraindications for spinal anesthesia
* skin lesions at injection site
* depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative cognitive disfunction | 6 months
  evaluated by Montreal Cognitive Assesment

SECONDARY OUTCOMES:
the influence of benzodiazepines on POCD | 6 months
  evaluated by Montreal Cognitive Assesment

CONTACTS AND LOCATIONS:
Locations (1):
- I Department of Anaesthesiology and Intensive Care, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No